CLINICAL TRIAL: NCT04290741
Title: Emergency Department Acupuncture for Acute Musculoskeletal Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Duke Endowment (Other); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00104140
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-03

CONDITIONS: Musculoskeletal Pain
Keywords: Acupuncture; Pain; Emergency Department
MeSH Terms: conditions — Musculoskeletal Pain; Pain; Emergencies | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auricular (Battlefield) Acupuncture (Experimental): Auricular acupuncture involves placement of needles based on battlefield acupuncture protocol which involves the placement of needles in up to 5 sites on each ear to treat pain.
  Interventions: Procedure: Auricular (Battlefield) Acupuncture
- Peripheral Acupuncture (Experimental): Peripheral acupuncture involves placement of needles in up to 30 specific sites in the head, neck, arms from the shoulders to the hands, and legs from the knees to the feet
  Interventions: Procedure: Peripheral Acupuncture
- Control (No Intervention): Standard of care without acupuncture

INTERVENTIONS:
Procedure: Auricular (Battlefield) Acupuncture — Placement of needles based on battlefield acupuncture protocol which includes up to 5 sites on each ear to treat pain.
  Arms: Auricular (Battlefield) Acupuncture
Procedure: Peripheral Acupuncture — Placement of needles in up to 30 specific sites in the head, neck, arms from the shoulders to the hands, and legs from the knees to the feet
  Arms: Peripheral Acupuncture

SUMMARY:
The purpose of this project is to determine the feasibility, acceptability and effectiveness of acupuncture in the Emergency Department (ED) for treating acute musculoskeletal pain. The overall goal is to reduce acute and subacute opioid use by improving acute pain, anxiety and disability with non-pharmacologic treatment options at a critical entry point for patients into the healthcare system. This full-scale randomized controlled trial (RCT) has been statistically powered to test the effectiveness of ED-based acupuncture for both one-hour (Stage 1) and one-month (Stage 2) pain reduction outcomes. The feasibility will be assessed based on patient recruitment and retention rates, while the acceptability will be assessed using patient reported outcomes and qualitative semi-structured interviews.

Stage 1 is a 2-phase study design. Phase (1): Enrolled subjects will be randomized to auricular (ear) acupuncture, peripheral acupuncture, or the control group receiving no acupuncture. Subjects assigned to an acupuncture arm will receive information and access to acupuncture in an outpatient clinic for the 4 weeks following ED visit. Subjects may also have a blood draw for biomarker analysis during their ED visit. A planned interim analysis of the first 60 patients (2/3 of the Phase 1 arm completed) will be completed to select the more effective and/or acceptable arm for Phase 2. At interim analysis, it was determined by the DSMB that neither arm was superior, so the recommendation was to continue Stage 1 Phase 2 unchanged with 3 arms. Stage 1 is complete, and we will proceed with Stage 2 powered to the 4-week pain score outcome. Stage 2 will proceed with the same procedures as stage 1, only powered to a different outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Clinical diagnosis of acute (≤7 days) musculoskeletal pain as determined by an ED provider
* Able to read and understand the consent form in English

Exclusion Criteria:

* Unable to receive acupuncture due to injury or infection of acupuncture sites
* Unwilling or unable to attend the follow-up outpatient acupuncture clinic
* Severe hearing or speech impairment
* Cognitive impairment, including evidence of drug, medication or alcohol intoxication, that would prevent comprehension of consent procedures or study measures and procedures
* Critical illness
* Deformity
* Medical condition that would contraindicate safe participation as determine by an ED provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score | ED pre-acupuncture (baseline); ED post-acupuncture (up to 1 hour); 2 and 4 weeks post discharge
  11-point Numeric Rating Scale (NRS) for current pain
Number of ED patients eligible for recruitment as measured by patient log | Post implementation, up to 6 weeks
Number of patients enrolled as measured by patient log | Post implementation, up to 6 weeks
Number of patients retained in study as measured by patient log | Post implementation, up to 6 weeks
Number of patients that found acupuncture satisfactory via satisfactory questionnaire | Post implementation, up to 6 weeks
  Likert-scale, agree disagree
Number of outpatient acupuncture sessions attended | 4 weeks post discharge
Number of adverse events | Post implementation, up to 2 weeks

SECONDARY OUTCOMES:
Change in function | ED pre-acupuncture (baseline); ED post-acupuncture (up to 1 hour); 2 and 4 weeks post discharge
  PROMIS-29
Change in cognitive function | ED pre-acupuncture (baseline); ED post-acupuncture (up to 1 hour); 2 and 4 weeks post discharge
  Neuro-QoL
Number of return ED visits | Up to one year post ED visit
Pain medications received | Up to three months post ED visit
Time in minutes for ED based acupuncture session | Post ED acupuncture session, up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Eucker, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital Emergency Department, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eucker SA, Glass O, Staton CA, Knisely MR, O'Regan A, De Larco C, Mill M, Dixon A, TumSuden O, Walker E, Dalton JC, Limkakeng A, Maxwell AMW, Gordee A, Kuchibhatla M, Chow S. Acupuncture for acute musculoskeletal pain management in the emergency department and continuity clinic: a protocol for an adaptive pragmatic randomised controlled trial. BMJ Open. 2022 Sep 23;12(9):e061661. doi: 10.1136/bmjopen-2022-061661. PMID 36153034

DOCUMENTS (1):
  • Informed Consent Form (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT04290741/ICF_000.pdf